CLINICAL TRIAL: NCT03616977
Title: Bioequivalence Study Comparing 2 Formulations of LY900014 in Healthy Subjects
Brief Title: Study to Compare 2 Formulations of LY900014 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 17152; I8B-MC-ITSS (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-08-01; First posted 2018-08-06 (Actual); Results first posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2018-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LY900014 U-200 (Experimental): Single subcutaneous (SC) dose of LY900014 U-200 in two of four study periods.
  Interventions: Drug: LY900014 U-200
- LY900014 U-100 (Experimental): Single SC dose of LY900014 U-100 in two of four study periods.
  Interventions: Drug: LY900014 U-100

INTERVENTIONS:
Drug: LY900014 U-200 — Administered SC
  Other Names: Ultra-Rapid Lispro
  Arms: LY900014 U-200
Drug: LY900014 U-100 — Administered SC
  Other Names: Ultra-Rapid Lispro
  Arms: LY900014 U-100

SUMMARY:
The study involves a comparison of 2 formulations of LY900014, which is a type of fast acting insulin. Study participants will be administered LY900014 U-100 two times and LY900014 U-200 two times, over 4 study periods, by injection under the skin. Blood samples will be taken to compare how the body handles the study drugs and how they affect the blood sugar levels. Side effects and tolerability will be documented. The study will last about 4 weeks, not including screening and follow up. Screening is required within 28 days prior to the start of the study and follow up is required at least 2 weeks after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

- Healthy male or a female (not pregnant and agreeable to take birth control measures until study completion)

* Have a body mass index (BMI) of 18 to 30 kilogram per square meter (kg/m²)
* Have normal blood pressure, pulse rate, electrocardiogram (ECG), blood and urine laboratory test results that are acceptable for the study
* Have veins suitable for easy blood collection and glucose solution infusion

Exclusion Criteria:

- Are currently participating in or completed a clinical trial within the last 30 days or any other type of medical research judged to be incompatible with this study

* Had donated blood of more than 450 milliliters (mL) or participated in a clinical trial with similar blood loss within the last 3 months
* Have a regular alcohol intake greater than 21 units/week (male), or 14 units/week (female)
* Smoke more than 10 cigarettes per day
* Are infected with hepatitis B or human immunodeficiency virus (HIV)
* Are taking illegal drugs

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2018-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

REFERENCES:
- [Derived] Linnebjerg H, LaBell ES, Dellva MA, Coutant DE, Leohr J. Bioequivalence of Ultra Rapid Lispro (URLi) U100 and U200 Formulations in Healthy Subjects. Diabetes Ther. 2020 Aug;11(8):1709-1720. doi: 10.1007/s13300-020-00848-4. Epub 2020 Jun 13. PMID 32535742

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Single SC dose of LY900014 U-200 in Periods 1 and 3. Single SC dose of LY900014 U-100 in Periods 2 and 4.
- Sequence 2: Single SC dose of LY900014 U-100 in Periods 1 and 3. Single SC dose of LY900014 U-200 in Periods 2 and 4.
Period: Period 1
Arm/Group | Sequence 1 | Sequence 2
Started | 34 | 35
Received at Least One Dose of Study Drug | 34 | 34
Completed | 34 | 34
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1
Period: Period 2
Arm/Group | Sequence 1 | Sequence 2
Started | 34 | 34
Completed | 34 | 34
Not Completed | 0 | 0
Period: Period 3
Arm/Group | Sequence 1 | Sequence 2
Started | 34 | 33 (Participant completed Period 2 and withdrew from the study.)
Received Study Drug | 33 (Participant not dosed due to adverse event.) | 32 (Participant not dosed due to adverse event.)
Completed | 33 | 32
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1
Period: Period 4
Arm/Group | Sequence 1 | Sequence 2
Started | 33 | 32
Completed | 33 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Overall: Single subcutaneous (SC) dose of LY900014 U-200 in two of four study periods. Single SC dose of LY900014 U-100 in two of four study periods.
Arm/Group | Overall
Number analyzed (Participants) | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 67
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 68
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 67
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 68

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Insulin Lispro Area Under the Concentration Curve From Time Zero to 10 Hours(h) (AUC [0-10h]) Following Administration of Each Study Arm
Description: Pharmacokinetics (PK): Insulin Lispro AUC time zero to 10 hours.
Time Frame: Period 1 through 4 Day 1: Predose, 5 minutes(m),10m,15m, 20m, 25m, 30m, 35m, 40m, 45m, 50m, 55m, 60m, 70m, 90m, 120m,150m,180m, 240m, 300m, 360m, 420m, 480m, 540m, and 600m postdose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomole times hour per liter (pmol*h/L)
Arm/Group | LY900014 U-100 | LY900014 U-200
Number analyzed (Participants) | 68 | 68
picomole times hour per liter (pmol*h/L) | 1690 (18) | 1710 (17)
Statistical Analysis 1: Comparison: LY900014 U-100 vs LY900014 U-200; Test type: Equivalence — Bioequivalence will be concluded if the 2-sided 90% Confidence Interval is completely contained within the interval (0.80, 1.25); Ratio of geometric least squares means = 1.01, 90% CI 2-sided [0.961 to 1.06]

2. Secondary Outcome: Glucodynamics (GD): Total Amount of Glucose Infused (Gtot) Over Duration of Clamp Following Administration of Each Study Arm
Description: GD: Gtot is the total glucose infusion over the clamp duration (10 hours) and is used to measure the study drug action over time as measured by the euglycemic clamp procedure. During the euglycemic clamp procedure, blood glucose concentrations are held constant after the administration of study treatment by adjusting the exogenous glucose infusion rate.
Time Frame: Period 1 through 4 Day 1: Predose, every 10 minutes(m) for 30m prior to dosing; During clamp: every 2.5m for 30m; every 5m for 30 to 120m; every 10m for 120 to 480m, and every 20m for 480m to 600m postdose
Population: All participants who received at least one dose of study drug and have evaluable glucodynamic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligram per kilogram (mg/kg)
Groups:
- LY900014 U-200: Single SC dose of LY900014 U-200 in two of four study periods.
  LY900014 U-200: Administered SC
Arm/Group | LY900014 U-100 | LY900014 U-200
Number analyzed (Participants) | 68 | 68
milligram per kilogram (mg/kg) | 1530 (46) | 1620 (45)

ADVERSE EVENTS:
Time Frame: Baseline to end of study (Up to 62 days)
Description: All participants who received at least one dose of study drug.
Groups:
- LY900014 U-100: Single SC dose of LY900014 U-100.
- LY900014 U-200: Single SC dose of LY900014 U-200.
Arm/Group | LY900014 U-100 | LY900014 U-200
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/68
Other Adverse Events (participants affected / at risk) | 20/68 | 19/68
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY900014 U-100 (N=68) | LY900014 U-200 (N=68)
Catheter site swelling (General disorders) | 4 (5) | 0 (0)
Infusion site pain (General disorders) | 4 (4) | 3 (4)
Infusion site swelling (General disorders) | 10 (10) | 10 (10)
Headache (Nervous system disorders) | 7 (8) | 7 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-07-20): https://cdn.clinicaltrials.gov/large-docs/77/NCT03616977/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/77/NCT03616977/SAP_001.pdf